CLINICAL TRIAL: NCT03153007
Title: Qualitative Research in Patients With Diabetic Foot Ulcer
Brief Title: Study of Subjects With Diabetic Foot Ulcer (DFU)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: 207650
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with DFU: Adult male or female subjects, 18 years of age or over and currently receiving treatment for a diagnosis of DFU or have received treatment for a past foot ulcer within the last 6 months, will be recruited from up to three clinical sites. They will undergo concept elicitation interviews over the telephone or in-person by trained and experienced interviewers.

SUMMARY:
Foot ulceration is a common and costly complication of diabetes. GSK1278863 is a topical drug, which is being developed to treat wounds associated with DFU. The aim of this study is to explore the symptoms and impacts of DFU from the subject perspective and to elicit in-depth information about DFU signs and symptoms, impacts on functioning and health-related quality of life (HRQoL). Adult DFU subjects with current or recent (within last six months) neuropathic foot ulcers will be eligible to participate in this prospective, cross-sectional interview study. Approximately 20 DFU subjects will be recruited from up to three clinical sites. Potential subjects will be pre-screened and then contacted to gauge interest in the study. Interested subjects will be screened and eligible subjects will consent to release contact information to research staff. Research staff will contact the subject to schedule interviews. This study will include concept elicitation interviews over the telephone or in-person by trained and experienced interviewers. In-person interviews will be conducted in a private room at the clinical site. All interviews will be conducted in English and will be guided by semi-structured interview guides. All subjects will provide written consent prior to the start of the interview.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 18 years of age or over
* Has a diagnosis of type 1 or 2 diabetes
* Has a diagnosis of neuropathic foot ulcer with minimal, if any, ischemia present (Ankle-Brachial Index [ABI] >=0.6 or transcutaneous oxygen [TcPO2] >35 millimeter of mercury [mmHg])
* Wagner grade 1 or 2
* Currently receiving treatment for a diagnosis of diabetic foot ulcer or have had an active foot ulcer healed within the last 6 months
* Is not currently enrolled in a clinical trial for DFU
* Is willing and able to provide informed consent indicating that they understand the purpose and procedures required for the study
* Is willing and able to participate in the study which includes a 60 minute interview
* Willing to have interview audio-recorded
* Speaks English as primary language

Exclusion Criteria:

* Subjects who does not meet the inclusion criteria
* Has diagnosis of critical limb ischemia
* Has ulcers that have exposure of tendon, bone, or joint capsule (Wagner grade >2)
* Has osteomyelitis or gangrenous ulcers
* Is currently enrolled in a clinical trial for DFU
* Is unwilling or unable to sign an informed consent document indicating that they understand the purpose and procedures of the study
* Is unwilling or unable to participate in the study which includes an interview of up to 60 minutes in duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 20 DFU adult male or female subjects, 18 years of age or over, with current or recent (within last six months) neuropathic foot ulcers will be recruited from up to three clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Assessment of signs and symptoms, impacts on functioning and HRQoL among subjects with DFU | Up to 60 minutes
  An iterative and thematic analytic approach will be applied to the concept elicitation data in order to identify key concepts related to DFU signs and symptoms, impacts on functioning and HRQoL. Concepts that emerge from the analysis will be tracked using a saturation matrix and will be recorded until saturation is attained, or at the point when no new concepts have emerged from the data. Transcripts produced from the subject and expert interview audio recordings will be analyzed using qualitative analysis software in order to identify themes emerging from the data while accounting for information gleaned from the review of literature.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bethesda, Maryland, United States

REFERENCES:
- See also: Results for study 207650 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/207650?search=study&search_terms=207650#rs